CLINICAL TRIAL: NCT03140995
Title: Does Exercise Have an Impact on Sleep and Mood in People Who Have Rheumatoid Arthritis: a Pilot Randomised Controlled Trial
Brief Title: Sleep and Exercise in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Limerick (Other)
Collaborators: University of Limerick (Other)
Responsible Party: Principal Investigator, Sean McKenna, PhD Candidate, University Hospital of Limerick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GOIPG/2016/58
Record Dates: First submitted 2017-04-25; First posted 2017-05-04 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Rheumatoid Arthritis; Inflammatory Arthritis
Keywords: Exercise; Sleep
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single centre, single blinded pilot randomised controlled trial, comparing an aerobic intermittent exercise training intervention (walking programme) against verbal and written instructions regarding the benefits of exercise in RA.
Who Masked: Outcomes Assessor
Masking Description: At baseline assessment demographic information and outcome measures will be collected by a physiotherapist not involved in the intervention and will be blinded to which arm the participant has been allocated to. This will all take place at the Department of Clinical Therapies, University of Limerick.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Active Comparator): The walking programme will consist of a total of 21 aerobic walking sessions, with 1 per week being supervised by a trained physiotherapist, spread over a maximum of eight weeks (2-3 times/week). During the first 4 weeks the intention is to increase frequency and the final 4 weeks the intensity, using the Borg Rate of Perceived exertion 6-20 or distance from 2km to 6km. The participants will attend the University of Limerick for a final assessment at week 9.
  Interventions: Behavioral: Walking Programme
- Control Group (No Intervention): The control group will be given verbal and written instructions regarding the benefits of exercise in RA.

INTERVENTIONS:
Behavioral: Walking Programme — The programme will be devised using incremental targets for daily walks based on the 6-20 Borg of rating of perceived exertion scale (Borg RPE). They will be instructed that they should be moderately short of breath on exertion i.e. unable to comfortably hold a conversation while walking
  Arms: Exercise Intervention

SUMMARY:
Regular physical activity is important for people with rheumatoid arthritis (RA). Sleep requirements for adults should be on a 'sleep needs spectrum' of between 7 to 9 hours per day. Poor sleep is a common complaint among people with RA, which may have an effect on their activity levels and well-being. There is evidence that physical activity and exercise can improve sleep quality and disturbances in other chronic disease populations therefore, examining how same affects sleep in RA is important.

DETAILED DESCRIPTION:
Sleep is an important aspect in maintaining the body's circadian rhythm. In general getting fewer than 5 hours sleep per day has been associated with cardiovascular problems, diabetes and obesity and can also be linked to depression and anxiety. Poor sleep is a common complaint among people with rheumatoid arthritis (RA) with disturbed sleep and fatigue known to affect up to 70% in this population. Poor sleep quality may contribute to the feelings of pain, fatigue and poor psychological well-being which in turn may further deteriorate functional ability and reduced activity.

It is known that exercise improves a person's psychological state which can also be an additional factor in improving or indeed disrupting quality of sleep. Exercise has been identified as an important part of the nonpharmacological management of poor sleep and in improving sleep quality however, people with RA were previously cautioned about undertaking exercise. Therefore, changes in sleep quality during exercise intervention should be evaluated so that society can understand more the potential for long-term changes in overall health status, in people who have RA. Indeed the intensity level of the activity in people with RA may be of additional importance.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be eligible to participate if they are aged 18-70; have a diagnosis of RA (defined by the American College of Rheumatology 1987 criteria); have poor sleep (Pittsburgh Sleep Quality Index global score >5); have a low disease score on 28 joints (DAS28) <3.2; Health Assessment Questionnaire result of <2.4 and are able to provided informed consent, understand and speak English. All the above will be determined should the person be interested in participating and before any fitness testing will be place.

Exclusion Criteria:

* Participants will be excluded from the study if they have severe physical disability (HAQ score > 2.5); are pregnant; participate in regular physical activity in their leisure time (self-reported aerobic exercise > 5 times per week); have cardiac symptoms corresponding to New York Heart Association (NYHA) functional classification > 2;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 8 Weeks
  Sleep

SECONDARY OUTCOMES:
RA related Pain - visual analog scale (VAS) consisting of a 10cm horizontal line anchored from 0 (no pain) to 10 (worst pain possible). | up to 8 weeks follow up
  Pain
Profile of Moods State | up to 8 weeks
  Mood
Quick Inventory of Depressive Symptomatology | up to 8 weeks
  Depression
State Trait Anxiety Inventory | up to 8 weeks
  Anxiety
Health Assessment disability Index | up to 8 weeks
  Functional limitation
Disease Activity Score with 28 joints | up to 8 weeks
  Disease activity
Rheumatoid Arthritis-Specific Quality of Life Instrument | up to 8 weeks
  Quality of Life
Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaire | up to 8 weeks
  Fatigue
Exercise Benefits and Barriers Scale | up to 8 weeks
  Exercise barriers

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Limerick, Limerick, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Yes
The investigating team only will have access to the patient's names and/or identifying factors for participants at the site and University of Limerick (UL) researchers will have access to the full data set from the single site. Participants will be allocated a study code. Thereafter It is anticipated that the results will be used in presentations to conferences such as European League against Rheumatism (EULAR) and American College of Rheumatology (ACR). Additionally papers will be prepared for submission to peer reviewed journals, through Arthritis Ireland and the UL Research office. Results will also be made available at aggregate level to Consultant Rheumatologists Dr. Alexander Fraser and Dr. Joe Devlin, Department of Rheumatology, University Hospitals Limerick. Results will be shared via supplementary material thereafter.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Early 2020

REFERENCES:
- [Result] McKenna S, Donnelly A, Fraser A, Comber L, Kennedy N. Does exercise impact on sleep for people who have rheumatoid arthritis? A systematic review. Rheumatol Int. 2017 Jun;37(6):963-974. doi: 10.1007/s00296-017-3681-x. Epub 2017 Mar 1. PMID 28251248
- [Result] McKenna S, Donnelly A, Fraser A, Kennedy N. Sleep and physical activity: a survey of people with inflammatory arthritis and their engagement by health professionals in rheumatology in Ireland. Disabil Rehabil. 2018 Sep;40(19):2260-2266. doi: 10.1080/09638288.2017.1334095. Epub 2017 Jun 2. PMID 28573870
- [Result] McKenna S, Tierney M, O'Neill A, Fraser A, Kennedy N. Sleep and physical activity: a cross-sectional objective profile of people with rheumatoid arthritis. Rheumatol Int. 2018 May;38(5):845-853. doi: 10.1007/s00296-018-4009-1. Epub 2018 Mar 14. PMID 29541902
- [Result] McKenna S, Kelly G, Kennedy N. A survey of physiotherapists' current management and the promotion of physical activity, in people with rheumatoid arthritis. Disabil Rehabil. 2019 Sep;41(18):2183-2191. doi: 10.1080/09638288.2018.1461258. Epub 2018 Apr 12. PMID 29644891
- [Result] McKenna SG, Donnelly AE, Esbensen BA, Fraser AD, Kennedy NM. The impact of exercise on sleep (time, quality, and disturbance) in patients with rheumatoid arthritis: a study protocol for a pilot randomised controlled trial. Rheumatol Int. 2018 Jul;38(7):1191-1198. doi: 10.1007/s00296-018-4052-y. Epub 2018 May 15. PMID 29766257
- [Derived] McKenna SG, Donnelly A, Esbensen BA, Comber L, Ng WL, Anjum AM, Fraser A, Kennedy NM. The feasibility of an exercise intervention to improve sleep (time, quality and disturbance) in people with rheumatoid arthritis: a pilot RCT. Rheumatol Int. 2021 Feb;41(2):297-310. doi: 10.1007/s00296-020-04760-9. Epub 2021 Jan 2. PMID 33386901
- See also: The impact of exercise on sleep (time, quality, and disturbance) in patients with rheumatoid arthritis: a study protocol for a pilot randomised controlled trial — https://link.springer.com/article/10.1007/s00296-018-4052-y